CLINICAL TRIAL: NCT05778201
Title: To Study the Effects of Baby Drink on Vision Care
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hui Wen Lin, Clinical Professor, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRREC-111-088
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Baby Drink Intervention group
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Baby Drink group (Experimental): 1 package/ day for 1 month
  Interventions: Biological: Baby Drink group

INTERVENTIONS:
Biological: Baby Drink group — 1 packge (20 ml)/ day for 1 month

SUMMARY:
Baby Drink is a formula based on lutein, mixed with blueberry fermented liquid, vitamins and minerals. Lutein is an effective antioxidant to prevent retinal damage caused by blue light, but it cannot be produced in the human body and depends on dietary intake. Blueberry fermented liquid is rich in polyphenolic compounds with excellent antioxidant capacity and the potential to reduce oxidative damage to eye cells caused by ultraviolet rays. With the prevalence of 3C products, myopia patients are increasing year by year in various regions, and suffer from eye diseases or vision loss with different degrees of complications. In this study, the subjects were provided with Baby Drink and tracked the degree of visual fatigue by regular questionnaires, and measured for visual acuity, axial length and diopter. The aim of this study is to investigate the protection of Baby Drink on visual acuity and visual fatigue.

DETAILED DESCRIPTION:
1. Visual acuity measurement: Snellen's Chart was used to measure visual acuity.
2. Refractive examination: Measure binocular refraction with Open Field computer refractor (Shin-Nippon Nvision K5001 Wide View).
3. Measuring the axial length of the eye: Use the multifunctional optical eyeball length measuring instrument (Lenstar) to measure the distance from the instrument to the optical paths such as the cornea, lens, and retina, and then convert to the axial length of the eye.
4. Corneal radian measurement: Use a keratometer (Bausch & Lomb Keratometer) to measure the corneal radian and curvature, and estimate the degree of corneal astigmatism.
5. Visual fatigue questionnaire survey: A visual fatigue scale questionnaire was designed using Ocular Surface Disease Index (OSDI) and Computer Vision Syndrome (CVS).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 or over
2. Willing to participate in this study and sign the subject's consent form
3. Myopia less than 700 degrees

Exclusion Criteria:

1. Have consumed related eye care products in past 3 months
2. Those who have eye infection in the past 3 months
3. People who have been diagnosed with any eye diseases in past 3 months
4. Those who are allergic to cicadae

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Eye fatigue questionnaire | 1 month
  1. Eye fatigue were evaluated according to The Ocular Surface Disease Index (OSDI) introduced in 1997 by the Outcomes Research Group (Allergan Inc., Irvine, CA).
  2. Content including: (1) Eye swelling, (2) Eye soreness, (3) Photophobia, (4) Blurred vision, (5) Dry eye, (6) Foreign body sensation, (7) Tearing, (8) General discomfort related to eye fatigue.
  3. Scores are expressed on a scale of 0-3. 0 = No symptoms , 1 = Occasionally (≤1 time/day), 2 = Sometimes (1-3 times/day), 3 = Frequently (>3 times/day), a low score means less visual fatigue and better eye quality.
Best vision test | 1 month
  1. Visual acuity was tested with the Snellen Eye Test Chart and recorded with the score proposed by Snellen.
  2. Subjects were asked to stand 20 feet away to observe the snellen E-chart and record the smallest visual mark.
  3. Recording method: 20/20 (1.0) is defined as normal vision, lower than this score indicates that the subject has ametropia, and higher than this indicates that the subject's vision is higher than the general standard

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wen Lin, ph.D, Principal Investigator — Asia University
Locations (1):
- Asia university, Taichung, Taiwan